CLINICAL TRIAL: NCT01090869
Title: Physical Activity is Healthy - Effect of Weight Loss or Physical Training Per se?
Brief Title: Physical Training Per se
Acronym: TPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Ph.D., D.Ms. Bente M. Stallknecht, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-KF-2006-6443
Record Dates: First submitted 2010-03-16; First posted 2010-03-23 (Estimated); Last update posted 2010-03-23 (Estimated); Status verified 2007-10

CONDITIONS: Insulin Sensitivity
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Physical training, unchanged diet (Active Comparator): Daily endurance training equivalent to 600 kcal/day and unchanged habitual diet
  Interventions: Behavioral: 12 weeks of lifestyle change
- Physical training, increased diet (Active Comparator): Daily endurance training equivalent to 600 kcal/day, and increased diet by 600 kcal/day.
  Interventions: Behavioral: 12 weeks of lifestyle change
- Diet, unchanged physical activity (Active Comparator): Energy-reduced diet by 600 kcal/day, and unchanged sedentary lifestyle
  Interventions: Behavioral: 12 weeks of lifestyle change
- Control (No Intervention): Unchanged sedentary lifestyle and diet
  Interventions: Behavioral: 12 weeks of lifestyle change

INTERVENTIONS:
Behavioral: 12 weeks of lifestyle change — Participants were randomly assigned to a 12-week intervention in one of four groups: Training (T), energy-reduced Diet (D), Training and increased- Diet (T-iD) or Control (C). The interventions consisted of: T: increased physical activity through daily endurance training equivalent to 600 kcal/day, unchanged diet; D: sedentary lifestyle, reduced diet by 600 kcal/day primarily through reducing serving sizes and substituting energy dense with less energy dense nutrients; T-iD: increased physical activity through daily endurance training equivalent to 600 kcal/day, increased diet by 600 kcal/day primarily through increasing serving sizes and consuming energy dense nutrients; C: sedentary lifestyle and unchanged diet.

SUMMARY:
The investigators aimed to evaluate the health benefits of physical training per se, weight loss per se and exercise-induced weight loss in young, overweight men. The investigators hypothesized that physical training would have independent effects on various health parameters (insulin sensitivity, fasting glucose and insulin, total and abdominal fat mass, waist circumference, blood pressure and key muscle proteins), and that a concomitant weight loss from physical activity would increase the effect.

DETAILED DESCRIPTION:
At baseline, during the intervention and in the week following the intervention participants underwent a panel of tests:

* Cardio respiratory fitness
* blood pressure
* anthropometric measures

At baseline and after the intervention a hyperinsulinemic, euglycemic clamp were performed to asses insulin sensitivity.

Tissue and blood samples were also collected for further analysis:

* Total-protein analysis of selected proteins
* Fasting plasma glucose, insulin and free fatty acids

ELIGIBILITY:
Inclusion Criteria:

* Overweight (body mass index 25-30 kg/m2)
* Weight stable (±2 kg during the past 6 months)
* Body fat% >25%,
* Maximal oxygen uptake <45 mL/min/kg
* Sedentary and healthy according to interview
* Fasting glucose <6.1 mmol/L
* Blood pressure <140/90 mmHg
* No first degree relatives with type-2-diabetes

Exclusion Criteria:

* Resistance training
* Inability to meet intervention criteria

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2007-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Change in insulin sensitivity | week 0 and 13
  Before and after the 12 week interventions a 1-step, 120 min, hyperinsulinaemic, euglycemic clamp was performed. After an initial 2mL bolus of insulin infusate, insulin was infused at 40 microU/min/kg.

SECONDARY OUTCOMES:
Changes in body composition | DEXA: week 0, 2, 6, 10, and 13; MRI: Week 0 and 13
  Before, during and after the 12-week interventions changes in: Body mass, Lean body mass, Fat mass, Abdominal fat mass, and Viceral and subcutaneous fat were assesed by DEXA and MRI scans.

CONTACTS AND LOCATIONS:
Overall Officials: Pernille Nordby, MSc, Principal Investigator — University of Copenhagen
Locations (1):
- University of Copenhagen, Faculty Of Health Sciences, Department of Biomedical Sciences, Copenhagen, Denmark